CLINICAL TRIAL: NCT01026974
Title: A Phase 2, Open-Label, Single-Center, Extension Study Evaluating Antibody Persistence Compared to Naïve Children and Safety, Tolerability and Immunogenicity of a Booster Dose of Novartis rMenB±OMV NZ Vaccine in Healthy UK Children Who Previously Received a Three-Dose Series of the Novartis Vaccine as Infants in Study V72P9
Brief Title: Extension Study Evaluating Antibody Persistence and Safety, Tolerability and Immunogenicity of a Booster Dose of Novartis rMenB±OMV NZ Vaccine in Healthy UK Children Who Previously Received Three Doses of the Same Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V72P9E1; EUDRACT 2009-013075-21
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Meningococcal Disease
Keywords: Children; Pre-school; Meningococcal disease; Prevention; Vaccination
MeSH Terms: conditions — Meningococcal Infections

ARMS (4):
- 4rMenB (Experimental): Subjects received three primary doses of rMenB vaccine (at the age of 6-8 months; 2 months after and at 12 months) in parent study (NCT00433914) and one booster dose of rMenB vaccine at 40 months of age in the present study.
  Interventions: Biological: rMenB
- 4rMenB+OMV NZ (Experimental): Subjects received three primary doses of rMenB+OMV NZ vaccine (at the age of 6-8months; 2 months after and at 12 months) in parent study (NCT00433914) and one booster dose of rMenB+OMV NZ vaccine at 40 months of age in the present study.
  Interventions: Biological: rMenB+OMV NZ
- Naive_4042 (Experimental): Vaccine-naive subjects who received two catch -up doses of rMenB+OMV NZ vaccine at 40 and 42 months of age in the present study.
  Interventions: Biological: rMenB+OMV NZ
- Naive_6062 (Experimental): Vaccine-naive subjects who received two catch-up doses of rMenB+OMV NZ vaccine at 60 and 62 months of age in the present study.
  Interventions: Biological: rMenB+OMV NZ

INTERVENTIONS:
Biological: rMenB
  Arms: 4rMenB
Biological: rMenB+OMV NZ
  Arms: 4rMenB+OMV NZ; Naive_4042; Naive_6062

SUMMARY:
The proposed study V72P9E1 is an Extension Study of V72P9. The objectives of this extension study will be to explore antibody persistence in children at approximately 40 months of age and to evaluate the safety, tolerability and immunogenicity of a booster dose of rMenB±OMV NZ administered to subjects at approximately 40 months of age. Antibody persistence will be subsequently measured at 18-20 months after these booster doses when the subjects are 60 months of age. Two groups of naïve subjects, aged approximately 40 and 60 months, will be recruited in the study to serve as a baseline comparator for assessing antibody persistence at these ages. These subjects will receive a two-dose catch-up regimen with rMenB+OMV NZ. Subjects who are enrolled at 40 months of age are offered DTaP/IPV and MMR vaccinations , if they have not already received these vaccines prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 40 to 44-months-old children, who participated and completed the study V72P9 (follow-on subjects)
* Healthy 40 to 44-months or 60 to 62-months-old children (naïve subjects)

Exclusion Criteria:

* Previous ascertained or suspected disease caused by N meningitidis
* History of severe allergic reaction after previous vaccinations or hypersensitivity to any vaccine component
* Any serious chronic or progressive disease
* Known or suspected impairment/ alteration of the immune system
* Receipt of, or intent to immunize with another vaccine, within 30 days prior and after vaccination with the investigational vaccines (within 14 days for licensed flu vaccines)

Ages: 40 Months to 62 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2010-02; Primary Completion 2010-09 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Vaccine Group, Center for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford, Oxford, United Kingdom

REFERENCES:
- [Background] McQuaid F, Snape MD, John TM, Kelly S, Robinson H, Houlden J, Voysey M, Toneatto D, Kitte C, Dull PM, Pollard AJ. Persistence of bactericidal antibodies to 5 years of age after immunization with serogroup B meningococcal vaccines at 6, 8, 12 and 40 months of age. Pediatr Infect Dis J. 2014 Jul;33(7):760-6. doi: 10.1097/INF.0000000000000327. PMID 24722351
- [Derived] Snape MD, Philip J, John TM, Robinson H, Kelly S, Gossger N, Yu LM, Kittel C, Toneatto D, Dull PM, Pollard AJ. Bactericidal antibody persistence 2 years after immunization with 2 investigational serogroup B meningococcal vaccines at 6, 8 and 12 months and immunogenicity of preschool booster doses: a follow-on study to a randomized clinical trial. Pediatr Infect Dis J. 2013 Oct;32(10):1116-21. doi: 10.1097/INF.0b013e31829cfff2. PMID 23958808

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from a single center.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- 4rMenB: Subjects received three primary doses of rMenB vaccine (at the age of 6-8 months; 2 months after and at 12 months) in parent study and one booster dose of rMenB vaccine at 40 months of age in the present study.
- 4rMenB+OMV NZ: Subjects received three primary doses of rMenB+OMV NZ vaccine (at the age of 6-8 months; 2 months after and at 12 months) in parent study and one booster dose of rMenB+OMV NZ vaccine at 40 months of age in the present study.
- Naive_4042: Vaccine-naive subjects who received two catch-up doses of rMenB+OMV NZ vaccine at 40 and 42 months of age in the present study.
Period: Overall Study
Arm/Group | 4rMenB | 4rMenB+OMV NZ | Naive_4042 | Naive_6062
Started | 16 | 14 | 41 | 49
Completed | 15 | 12 | 29 | 46
Not Completed | 1 | 2 | 12 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 7 | 2
Not completed — Lost to Follow-up | 1 | 1 | 4 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Inappropriate enrollment | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4rMenB | 4rMenB+OMV NZ | Naive_4042 | Naive_6062 | Total
Number analyzed (Participants) | 16 | 14 | 41 | 49 | 120
Age, Continuous [Mean (Standard Deviation); unit: months] | 42.8 (1.1) | 43.1 (0.9) | 41.7 (1.7) | 61.3 (0.7) | 50.0 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 22 | 21 | 62
  Male | 8 | 3 | 19 | 28 | 58

OUTCOME MEASURES:

1. Primary Outcome: Persistence of Serum Bactericidal Antibody Titers in Children (at 40 Months of Age), Twenty-eight Months After Completing Primary Vaccination.
Description: The geometric mean antibody titers (GMTs) against Neisseria meningitidis serogroup B in children (at 40 months of age); twenty-eight months after completion of primary vaccination with either rMenB or rMenB+OMV NZ vaccines, are compared with the GMTs in vaccine-naïve children.
Time Frame: 28 months after primary vaccination; Baseline for Naïve
Population: Modified Intention-to-treat (MITT) population was defined as enrolled subjects who actually received at least one vaccine dose,and provided at least one evaluable serum sample both before and after baseline.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 4rMenB | 4rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 15 | 14 | 40
Titers
  44/76-SL strain (N = 14,14,39) | 1.26 [0.9 to 1.76] | 2.55 [1.15 to 5.66] | 1.08 [0.97 to 1.2]
  5/99 strain (N = 14,14,40) | 41 [18 to 95] | 29 [18 to 47] | 1 [1 to 1]
  NZ98/254 strain (N = 15,14,39) | 1 [1 to 1] | 1.74 [0.91 to 3.33] | 1 [1 to 1]
  M10713 strain ( N = 14,14,40) | 3.6 [1.32 to 9.84] | 7.11 [3.61 to 14] | 4.82 [2.9 to 8]

2. Secondary Outcome: Serum Bactericidal Antibody Titers in Children After a Single Booster Dose of rMenB or rMenB+OMV NZ Vaccine Given at 40 Months of Age
Description: The serum bactericidal antibody response one month after a booster dose of rMenB or rMenB+OMV NZ vaccine was given to children at 40 months of age is compared with the antibody titers following one catch-up dose rMenB+OMV NZ vaccine given at 40 months to vaccine-naive subjects and reported as GMTs.
Time Frame: 1 month post booster /1 month post dose 1 for Naïve
Population: Analysis was done on MITT population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 4rMenB | 4rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 14 | 14 | 39
Titers
  44/76-SL strain (N = 13,14,39) | 100 [50 to 200] | 114 [59 to 222] | 8.89 [5.83 to 14]
  5/99 strain (N=14, 14, 39) | 1007 [445 to 2277] | 926 [432 to 1988] | 27 [16 to 44]
  NZ98/254 strain (N=14, 14, 39) | 2.15 [0.88 to 5.23] | 32 [14 to 71] | 1.91 [1.35 to 2.71]
  M10713 strain (N = 13,14,39) | 10 [3.43 to 30] | 23 [13 to 41] | 6.04 [3.73 to 9.79]

3. Primary Outcome: Percentage of Subjects With Persisting Serum Bactericidal Antibodies Titers ≥4, Twenty-eight Months After Completing Primary Vaccination.
Description: The percentages of subjects with persisting serum bactericidal antibodies (hSBA) titers ≥4, against N meningitidis serogroup B at 40 months of age; twenty-eight months after completion of primary vaccination with either rMenB or rMenB+OMV NZ as compared to the vaccine-naïve children are reported.
  The serum bactericidal antibodies directed against serogroup B meningococci, are measured by human complement Serum Bactericidal Assay (hSBA).
Time Frame: 28 months after primary vaccination; Baseline for Naïve
Population: Analysis was done on MITT population
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | 4rMenB | 4rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 15 | 14 | 40
percentages of subjects
  44/76-SL strain (N = 14,14,39) | 14 [2 to 43] | 36 [13 to 65] | 3 [0.065 to 13]
  5/99 strain (N = 14,14,40) | 93 [66 to 100] | 100 [77 to 100] | 0 [0 to 9]
  NZ98/254 strain (N = 15,14,39) | 0 [0 to 22] | 14 [2 to 43] | 0 [0 to 9]
  M10713 strain (N = 14,14,40) | 29 [8 to 58] | 79 [49 to 95] | 53 [36 to 68]

4. Primary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events After a Booster Dose of rMenB or rMenB+OMV NZ Vaccine at Forty Months of Age.
Description: The safety and tolerability of a single booster dose of rMenB or rMenB+OMV NZ vaccine in 40 month old children who had previously received three primary doses of the same vaccine as infants in parent study was assessed in terms of number of subjects with solicited local and systemic reactions following vaccination and compared to tolerability in vaccine-naive children who received 1st catch-up dose of rMenB+OMV NZ at 40 months of age.
Time Frame: Day 1 to Day 7 [after booster vaccination /post dose 1 for naive]
Population: Analysis was done on the Safety population- defined as all subjects who received at least one Men B vaccination and provided post-baseline safety data.
Measure: Number; unit: participants
Groups:
- 4rMenB: Subjects received three primary doses of rMenB vaccine (at the age of 6-8months; 2 months after and at 12 months) in parent study and one booster dose of rMenB vaccine at 40 months of age in the present study.
- 4rMenB+OMV NZ: Subjects received three primary doses of rMenB+OMV NZ vaccine (at the age of 6-8months; 2 months after and at 12 months) in parent study and one booster dose of rMenB+OMV NZ vaccine at 40 months of age in the present study.
Arm/Group | 4rMenB | 4rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 16 | 14 | 39
participants
  Local | 14 | 14 | 38
  Injection-site pain | 10 | 12 | 34
  Injection-site erythema | 13 | 14 | 36
  Injection-site swelling | 9 | 6 | 10
  Injection-site induration | 11 | 5 | 17
  Systemic | 12 | 11 | 30
  Change in eating habits | 5 | 5 | 13
  Sleepiness | 6 | 6 | 20
  Vomiting | 0 | 2 | 1
  Diarrhea | 2 | 1 | 2
  Irritability | 8 | 11 | 24
  Headache | 2 | 1 | 4
  Arthralgia | 2 | 3 | 9
  Rash | 2 | 1 | 2
  Fever (≥38°C) | 4 | 1 | 6
  Other | 6 | 10 | 21
  Temperature (≥40°C) | 0 | 0 | 1
  Antipyretic preventive medication used | 4 | 9 | 19
  Antipyretic treatment medication used | 3 | 1 | 5
  Medically attended fever | 0 | 0 | 0

5. Secondary Outcome: Percentage of Subjects With Serum Bactericidal Antibody Titers ≥4 After Receiving a Single Booster Dose of rMenB or rMenB+OMV NZ Vaccine at 40 Months of Age
Description: The percentages of subjects with hSBA titers ≥4 against N meningitidis serogroup B one month after receiving a single booster dose of rMenB or rMenB+OMV NZ vaccine at 40 months of age, is compared with hSBA response following one catch-up dose of rMenB+OMV NZ vaccine given at 40 months in vaccine-naive subjects.
Time Frame: 1 month post-booster/ 1 month post-dose 1 for Naïve
Population: Analysis was done on MITT population.
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | 4rMenB | 4rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 14 | 14 | 39
percentages of subjects
  44/76-SL strain (N = 13, 14, 39) | 100 [75 to 100] | 100 [77 to 100] | 72 [55 to 85]
  5/99 strain (N=14, 14, 39) | 100 [77 to 100] | 100 [77 to 100] | 87 [73 to 96]
  NZ98/254 strain (N=14, 14, 39) | 21 [5 to 51] | 93 [66 to 100] | 23 [11 to 39]
  M10713 strain (N = 13, 14, 39) | 69 [39 to 91] | 93 [66 to 100] | 62 [45 to 77]

6. Secondary Outcome: Percentage of Subjects With a 4-fold Increase in Antibody Titers After a Single Booster Dose of rMenB or rMenB+OMV NZ Vaccine Given at 40 Months of Age
Description: The percentages of subjects with four-fold increase in hSBA titers over baseline against N meningitidis serogroup B, one month after receiving a single booster dose of rMenB or rMenB+OMV NZ vaccine at 40 months of age, and compared with 4-fold increase in hSBA titers following one catch-up dose of rMenB+OMV NZ vaccine given at 40 months to vaccine-naive subjects.
  Baseline was defined as either the time that the (first) booster dose was given (i.e. at 40 months of age) or the time of the first vaccination (i.e. at 40 months of age for Naive_4042 group.
Time Frame: 1 month post booster / 1 month post dose 1 for Naïve
Population: Analysis was done on MITT population
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | 4rMenB | 4rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 13 | 14 | 38
percentages of subjects
  44/76-SL strain (N = 11,14,37) | 100 [72 to 100] | 93 [66 to 100] | 54 [37 to 71]
  5/99 strain (N = 12,14,38) | 100 [74 to 100] | 100 [77 to 100] | 76 [60 to 89]
  NZ98/254 strain (N = 13,14,37) | 23 [5 to 54] | 71 [42 to 92] | 11 [3 to 25]
  M10713 strain (N = 11,14,38) | 18 [2 to 52] | 36 [13 to 65] | 5 [1 to 18]

7. Secondary Outcome: Persistence of Serum Bactericidal Antibody Titers in Children (at 60 Months of Age), Twenty Months After Receiving a Booster Dose of rMenB or rMenB+OMV NZ Vaccine
Description: The persisting serum bactericidal antibody titers in children (at 60 months of age), twenty months after receiving a booster dose of either rMenB or rMenB+OMV NZ vaccine (at 40 months of age) is compared with the antibody titers in vaccine -naïve subjects of the same age and reported as GMTs.
Time Frame: 20 months post booster/ Baseline for Naïve
Population: Analysis was done on the MITT population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 4rMenB | 4rMenB+OMV NZ | Naive_6062
Number analyzed (Participants) | 14 | 14 | 46
Titers
  44/76-SL strain (N = 9,12,46) | 9.37 [2.47 to 36] | 4.69 [1.98 to 11] | 1.09 [0.96 to 1.25]
  5/99 strain (N = 9,11,46) | 334 [186 to 599] | 119 [56 to 252] | 1.17 [0.96 to 1.42]
  NZ98/254 strain (N = 10,12,46) | 1 [1 to 1] | 1.63 [0.86 to 3.08] | 1 [1 to 1]
  M10713 strain (N = 8,11,45) | 4.96 [1.03 to 24] | 5.51 [2.19 to 14] | 8.09 [5.13 to 13]

8. Secondary Outcome: Percentage of Subjects With Persisting Serum Bactericidal Antibody Titers ≥4, Twenty Months After a Single Booster Dose of rMenB or rMenB+OMV NZ Vaccine
Description: The percentage of subjects (60 months of age) with persisting hSBA titers ≥4, twenty months after receiving a booster dose of either rMenB or rMenB+OMV NZ vaccine (at 40 months of age) are compared with hSBA response in vaccine-naïve subjects of the same age.
Time Frame: 20 months post booster/ Baseline for Naïve
Population: This analysis was done on MITT population
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | 4rMenB | 4rMenB+OMV NZ | Naive_6062
Number analyzed (Participants) | 10 | 12 | 46
percentages of subjects
  44/76-SL strain (N = 9,12,46) | 67 [30 to 93] | 67 [35 to 90] | 4 [1 to 15]
  5/99 strain (N = 9,11,46) | 100 [66 to 100] | 100 [72 to 100] | 4 [1 to 15]
  NZ98/254 strain 10, 12, 46) | 0 [0 to 31] | 17 [2 to 48] | 0 [0 to 8]
  M10713 strain (N = 8,11,45) | 50 [16 to 84] | 45 [17 to 77] | 67 [51 to 80]

9. Secondary Outcome: Percentage of Subjects With Serum Bactericidal Antibody Titers ≥4 Following Two Doses of rMenB+OMV NZ Vaccine Given One Month Apart, Either at 40 or 60 Months of Age
Description: The percentage of subjects with hSBA titers ≥4 after two catch-up doses of rMenB+OMV NZ vaccine when given either at- 40 & 42 months or 60 & 62 months of age is reported.
Time Frame: 1 month post -vaccine dose two
Population: Analysis was done on MITT population
Measure: Number (95% Confidence Interval); unit: percentages
Arm/Group | Naive_4042 | Naive_6062
Number analyzed (Participants) | 31 | 35
percentages
  44/76-SL strain (N = 30,34) | 100 [88 to 100] | 100 [90 to 100]
  5/99 strain (N = 31,34) | 100 [89 to 100] | 100 [90 to 100]
  NZ98/254 strain (N=31, 35) | 90 [74 to 98] | 89 [73 to 97]
  M10713 strain (N = 29,33) | 72 [53 to 87] | 97 [84 to 100]

10. Secondary Outcome: Serum Bactericidal Antibody Titers in Children Following Two Doses of rMenB+OMV NZ Vaccine Given One Month Apart, Either at 40 or 60 Months of Age.
Description: The serum bactericidal antibody response in children after two catch-up doses of rMenB+OMV NZ vaccine when given either at- 40 & 42 months or 60 & 62 months of age are reported as GMTs.
Time Frame: 1 month post vaccine dose two
Population: Analysis was done on MITT population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Naive_4042 | Naive_6062
Number analyzed (Participants) | 31 | 35
Titers
  44/76-SL strain (N = 30,34) | 74 [57 to 94] | 83 [67 to 103]
  5/99 strain (N = 31,34) | 247 [188 to 323] | 331 [254 to 432]
  NZ98/254 strain (N = 30,35) | 16 [11 to 23] | 14 [9.81 to 21]
  M10713 strain (N = 29,33) | 8.91 [5.19 to 15] | 44 [33 to 57]

11. Secondary Outcome: Percentage of Subjects With a 4-fold Increase in Antibody Titers After Two Catch up Doses of rMenB+OMV NZ Vaccine Given One Month Apart Either at 40 or 60 Months of Age
Description: The percentages of subjects with four-fold increase in hSBA titers over baseline against N meningitidis serogroup B one month after receiving a two catch-up doses of rMenB+OMV NZ vaccine either at 40 & 42 months or 60 & 62 months of age.
Time Frame: 1 month post vaccine dose 2
Population: Analysis was done on MITT population
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | Naive_4042 | Naive_6062
Number analyzed (Participants) | 31 | 35
percentages of subjects
  44/76-SL strain (N = 29,34) | 100 [88 to 100] | 100 [90 to 100]
  5/99 strain (N = 31,34) | 100 [89 to 100] | 100 [90 to 100]
  NZ 98/254 strain (N = 30,35) | 73 [54 to 88] | 69 [51 to 83]
  M10713 strain (N = 29,32) | 24 [10 to 44] | 53 [35 to 71]

12. Secondary Outcome: Persistence of Serum Bactericidal Antibody Titers in Children (at 60 Months), Eighteen Months After Receiving Two Catch-up Doses of rMenB+OMV NZ Vaccine.
Description: The serum bactericidal antibody response in children at 60 months of age who had received two catch-up doses of rMenB+OMV NZ vaccine at- 40 & 42 months age is reported as GMTs.
Time Frame: 18 months post vaccine dose 2
Population: Analysis was done on the MITT population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Naive_4042
Number analyzed (Participants) | 24
Titers
  44/76-SL strain | 2.73 [1.54 to 4.84]
  5/99 strain | 24 [16 to 35]
  NZ98/254 strain | 1 [1 to 1]
  M10713 strain (N = 23) | 14 [6.78 to 27]

13. Secondary Outcome: Percentage of Subjects With Serum Bactericidal Antibody Titers ≥4, Eighteen Months After Receiving Two Catch-up Doses of rMenB+OMV NZ Vaccine.
Description: Persisting hSBA titers ≥4 in children at 60 months of age, who had received two catch-up doses of rMenB+OMV NZ vaccine at 40 & 42 months age is reported.
Time Frame: 18 months post vaccine dose two
Population: Analysis was done on MITT population
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | Naive_4042
Number analyzed (Participants) | 24
percentages of subjects
  44/76-SL strain | 38 [19 to 59]
  5/99 strain | 100 [86 to 100]
  NZ98/254 strain | 0 [0 to 14]
  M10713 strain (N = 23) | 83 [61 to 95]

14. Secondary Outcome: Geometric Mean Antibody Concentrations in Children (at 40 Months of Age), Twenty Eight Months After Completing Primary Vaccination.
Description: The persisting geometric mean antibody concentrations (GMCs) against vaccine antigen 287-953 in children (at 40 months of age), twenty-eight months after completion of primary vaccination with either rMenB or rMen+OMV NZ vaccines, are compared with the GMCs in vaccine-naïve children.
  GMCs against vaccine antigen 287-953 were measured using enzyme linked immunosorbent assay (ELISA).
Time Frame: 28 months after primary vaccination/ Baseline for Naïve
Population: Analysis was done on MITT population.
Measure: Geometric Mean (95% Confidence Interval); unit: concentrations (AU/mL)
Arm/Group | 4rMenB | 4rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 14 | 14 | 39
concentrations (AU/mL) | 86 [43 to 173] | 103 [61 to 174] | 27 [22 to 35]

15. Secondary Outcome: Geometric Mean Antibody Concentrations in Children, After a Single Booster Dose of rMenB or rMenB+OMV NZ Vaccine Given at 40 Months of Age.
Description: The GMCs against vaccine antigen 287-953, in children one month after receiving a single booster dose of either rMenB or rMen+OMV NZ vaccine , is compared with GMCs following one catch-up dose of rMenB+ OMV NZ in children at 40 months.
Time Frame: 1 month post booster /1 month post dose 1 for Naïve
Population: Analysis was done on MITT population
Measure: Geometric Mean (95% Confidence Interval); unit: concentrations (AU/mL)
Arm/Group | 4rMenB | 4rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 15 | 14 | 39
concentrations (AU/mL) | 5187 [2924 to 9204] | 3662 [2065 to 6491] | 83 [52 to 133]

16. Secondary Outcome: Geometric Mean Antibody Concentrations in Children (at 60 Months of Age), Twenty Months After Receiving a Booster Dose of rMenB or rMenB+OMV NZ Vaccine
Description: The persisting GMCs against vaccine antigen 287-953 in children (at 60 months of age), twenty months after receiving a booster dose of either rMenB or rMenB+OMV NZ vaccine (at 40 months), are compared with GMCs in vaccine-naïve children of same age.
Time Frame: 20 months post booster/ Baseline for Naïve
Population: Analysis was done on MITT population.
Measure: Geometric Mean (95% Confidence Interval); unit: concentrations (AU/mL)
Arm/Group | 4rMenB | 4rMenB+OMV NZ | Naive_6062
Number analyzed (Participants) | 10 | 12 | 46
concentrations (AU/mL) | 772 [395 to 1512] | 358 [201 to 640] | 25 [19 to 33]

17. Secondary Outcome: Geometric Mean Antibody Concentrations in Children After Two Doses of rMenB+OMV NZ Vaccine Given One Month Apart, Either at 40 Months or 60 Months of Age.
Description: The GMCs against vaccine antigen 287-953 in children after two catch-up doses of rMenB+OMV NZ vaccine when given either at 40- & 42- months or 60- & 62- months of age are reported.
Time Frame: 1 month post vaccine dose two
Population: Analysis was done on the MITT population.
Measure: Geometric Mean (95% Confidence Interval); unit: concentrations (AU/mL)
Arm/Group | Naive_4042 | Naive_6062
Number analyzed (Participants) | 31 | 35
concentrations (AU/mL) | 612 [329 to 1139] | 2164 [1663 to 2817]

18. Secondary Outcome: Geometric Mean Antibody Concentrations in Children (at 60 Months), Eighteen Months After Receiving Two Catch-up Doses of rMenB+OMV NZ Vaccine.
Description: Persistence of GMCs against vaccine antigen 287-953 in children (60 months of age), eighteen months after two catch-up doses of rMenB+OMV NZ vaccine given at 40 months of age.
Time Frame: 18 months post vaccine dose 2
Population: Analysis was done on MITT population
Measure: Geometric Mean (95% Confidence Interval); unit: concentrations (AU/mL)
Arm/Group | Naive_4042
Number analyzed (Participants) | 24
concentrations (AU/mL) | 87 [63 to 120]

19. Secondary Outcome: Percentage of Subjects With Four Fold Increase in Geometric Mean Antibody Concentrations , After a Single Booster Dose of rMenB or rMenB+OMV NZ Vaccine Given at 40 Months of Age
Description: The percentage of subjects with four fold increase in GMCs over baseline against vaccine antigen 287-953 one month after receiving a single booster dose of either rMenB or rMen+OMV NZ vaccine, is compared with responses following one catch-up dose of rMenB+OMV NZ in children at 40 months.
Time Frame: 1 month post booster / 1 month post dose 1
Population: Analysis was done on MITT population
Measure: Number (95% Confidence Interval); unit: percentages of subjects
Arm/Group | 4rMenB | 4rMenB+OMV NZ | Naive_4042
Number analyzed (Participants) | 14 | 14 | 38
percentages of subjects | 100 [77 to 100] | 100 [77 to 100] | 21 [10 to 37]

20. Secondary Outcome: Percentage of Subjects With 4-fold Increase in Geometric Mean Antibody Concentrations, After Two Catch-up Doses of rMenB+OMV NZ Vaccine Given One Month Apart Either at 40 or 60 Months of Age
Description: The percentages of subjects with four-fold increase in GMCs over baseline against vaccine antigen 287-953, one month after receiving a two catch-up doses of rMenB+OMV NZ vaccine either at 40 & 42 months or 60 & 62 months of age.
Time Frame: 1 month post dose 2
Population: Analysis was done on MITT population
Measure: Geometric Mean (95% Confidence Interval); unit: percentages of subjects
Arm/Group | Naive_4042 | Naive_6062
Number analyzed (Participants) | 31 | 35
percentages of subjects | 77 [59 to 90] | 97 [85 to 100]

21. Secondary Outcome: Number of Children Reporting Solicited Local and Systemic Adverse Events After Receiving Two Catch-up Doses of rMenB+OMV NZ Vaccine One Month Apart, Either at 40 or 60 Months of Age
Description: The safety and tolerability of a two doses of rMenB+OMV NZ vaccine in children when given either at 40 & 42 months or 60 & 62 months of age is assessed in terms of number of subjects with solicited local and systemic reactions following vaccination.
Time Frame: Day 1-7 after each vaccination
Population: Analysis was done on the Safety population
Measure: Number; unit: participants
Arm/Group | Naive_4042 | Naive_6062
Number analyzed (Participants) | 39 | 48
participants
  Local | 39 | 48
  Injection-site pain | 38 | 46
  Injection-site erythema | 38 | 46
  Injection-site swelling | 19 | 32
  Injection-site induration | 26 | 28
  Systemic | 39 | 48
  Change in eating habits | 20 | 15
  Sleepiness | 26 | 26
  Vomiting | 4 | 7
  Diarrhea | 4 | 4
  Irritability | 29 | 29
  Headache | 8 | 12
  Arthralgia | 13 | 24
  Rash | 3 | 5
  Fever (≥38°C) | 10 | 10
  Other | 21 | 26
  Antipyretic Preventive medication used | 24 | 29
  Antipyretic Treatment medication used | 8 | 12
  Temperature(≥40°C) | 1 | 0
  Medically attended fever | 1 | 0

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected from Day 1 to Day 7 after each vaccination, SAEs and other unsolicited AEs were collected throughout the study [approximately 20 months for Groups rMenB; rMenB+OMV NZ and Naive_4042 and Days 1-91 for Naive_6062 group].
Description: The population reported in this section is the safety population.
Arm/Group | 4rMenB | 4rMenB+OMV NZ | Naive_4042 | Naive_6062
Serious Adverse Events (participants affected / at risk) | 1/16 | 1/14 | 4/41 | 1/48
Other Adverse Events (participants affected / at risk) | 15/16 | 14/14 | 41/41 | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 4rMenB (N=16) | 4rMenB+OMV NZ (N=14) | Naive_4042 (N=41) | Naive_6062 (N=48)
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Encephalitis (Nervous system disorders) | 0 | 0 | 1 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 4rMenB (N=16) | 4rMenB+OMV NZ (N=14) | Naive_4042 (N=41) | Naive_6062 (N=48)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 4 | 4
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 6 | 7
Injection site erythema (General disorders) | 13 | 14 | 40 | 46
Injection site induration (General disorders) | 11 | 5 | 26 | 28
Injection site pain (General disorders) | 10 | 12 | 38 | 46
Injection site swelling (General disorders) | 9 | 6 | 20 | 32
Irritability (General disorders) | 8 | 11 | 29 | 29
Pain (General disorders) | 1 | 0 | 1 | 0
Pyrexia (General disorders) | 4 | 1 | 11 | 10
Swelling (General disorders) | 2 | 1 | 0 | 0
Ear infection (Infections and infestations) | 2 | 1 | 3 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 3 | 2
Tonsillitis (Infections and infestations) | 0 | 1 | 4 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Varicella (Infections and infestations) | 1 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 13 | 24
Hair follicle tumor benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 8 | 13
Somnolence (Nervous system disorders) | 6 | 6 | 26 | 26
Eating disorder (Psychiatric disorders) | 5 | 5 | 20 | 15
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 5 | 5
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Ear tube insertion (Surgical and medical procedures) | 0 | 1 | 0 | 0
Induration (General disorders) | 0 | 1 | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days